CLINICAL TRIAL: NCT06136949
Title: The Theranostic Value of STARD3 in Colorectal Cancer: The STAR Study: a Monocentric Observational Study
Brief Title: The Theranostic Value of STARD3 in Colorectal Cancer: The STAR Study
Acronym: STAR
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2023-14
Record Dates: First submitted 2023-10-30; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at verifying the overexpression of STARD3 in both early and advanced CRC patients derived tissues, to identify the pathways underpinning tumorigenesis and cancer progression in which STARD3 is involved. Moreover its role as a dynamic biomarker of treatment response and its part in treatment sensitivity will be explored.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most prevalent and deadly tumours in both men and women worldwide. An RNAi screening on 214 potential oncogenes described by the TCGA was performed and STARD3 was identified as potential theranostic target in mCRC. Considering the effects on cell viability and the druggability, STARD3 represents a strong candidate as a valid diagnostic and therapeutic target for mCRC patients.

In recent years, organoids have become a research hotspot, showing a significant potential in the biological analysis of tumours. Patient derived organoids could be a viable platform to test clinically available drugs and/or promising new molecules to explore tumour sensitivity in an ex-vivo model.

This is a longitudinal observational study on CRC patients derived tissues to verify the overexpression of STARD3 in both early and advanced CRC patients, to identify the pathways underpinning tumorigenesis and cancer progression in which STARD3 is involved through the development of cancer derived organoids, to explore its role as a dynamic biomarker of treatment response and to demonstrate its part in treatment sensitivity measured in tumour derived organoids compared to drug sensitivity observed in real-world patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of colorectal cancer, independently from diagnosis stage.
* Age ≥18 years.
* Signed informed consent form.
* Availability of tissue and blood samples stored at the Institutional Biobank for research purposes.

Exclusion Criteria:

* Patients for which the tumour biobanking process could compromise the diagnostic assessments.
* Pregnancy or breast-feeding.
* History of concomitant or previous malignancy in the previous 5 years, except for adequately treated cutaneous squamous cell carcinoma or surgically removed in situ cervical carcinoma.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive CRC patients with available tumour tissue biopsies (primary surgery or diagnostic endoscopy) stored in the Institutional Biobank will be enrolled. Available biopsies collected from 1st January 2012 to 31st December 2027 will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of overexpression of STARD3 in both early and advanced CRC patients | at enrolment
  Frequency of STARD3 overexpression in both early and advanced CRC patients

SECONDARY OUTCOMES:
Frequencies of overexpression or downregulation of selected genes alteration related to STARD3 overexpression | up to 5 years
  Frequencies of overexpression or downregulation of selected genes alteration related to STARD3 overexpression. This analysis will be carried out in organoids cancer model
Presence of STARD3 overexpression as a prognostic factor | from enrolment to at least 5 years
  relation between presence of STARD3 overexpression (dichotomic variable) and disease-free survival (DFS) defined as time between enrollment and objective tumor progression using Kaplan Meyer method
Variation of STARD3 as a prognostic factor | from enrolment to at least 5 years
  STARD3 expression could change over the time and affect disease-free survival (DFS). Relation between variation of STARD3 overexpression (dichotomic variable) and DFS (defined as time between enrollment and objective tumor progression) will be accessed with Kaplan Meyer method.
Relation between presence of STARD3 overexpression and progression-free survival (PFS) | from enrolment to at least 5 years
  relation between presence of STARD3 overexpression (dichotomic variable) and progression-free survival (PFS) defined as time between enrollment and objective tumor progression or death whichever comes first, using Kaplan Meyer method
relation between variation of STARD3 overexpression and progression-free survival (PFS) | from enrolment to at least 5 years
  relation between variation of STARD3 overexpression (dichotomic variable) and progression-free survival (PFS) defined as time between enrollment and objective tumor progression or death whichever comes first, using Kaplan Meyer method
Relation between presence of STARD3 overexpression and Overall survival (OS | from enrolment to at least 5 years
  relation between presence of STARD3 overexpression (dichotomic variable) and Overall survival (OS) defined as time between enrollment and death, using Kaplan Meyer method
Relation between variation of STARD3 overexpression and Overall survival (OS) | from enrolment to at least 5 years
  Relation between variation of STARD3 overexpression (dichotomic variable) and Overall survival (OS) defined as time between enrollment and death, using Kaplan Meyer method
Difference in the mean variation of STARD3 level in patients receiving oncologic treatment, evaluated from start of treatment to the first revaluation and to disease progression | from enrolment to at least 5 years
  Difference in the mean variation of STARD3 level in patients receiving oncologic treatment, evaluated from start of treatment to the first revaluation and to disease progression
Demonstrate treatment sensitivity measured in tumour derived organoids | up to 5 years
  Description of IC50 value (inhibitory concentration 50) for each drug tested on tumour-derived organoids
Relation between treatment sensitivity measured in tumour derived organoids and treatment sensitivity in patients | up to 5 years
  Relation between IC50 (inhibitory concentration 50) calculated for each drug tested on patients' tumour-derived organoids and PFS of patients defined as time between enrollment and objective tumor progression or death whichever comes first. Relation will be measured with Hazard Ratio (HR)
Concordance between the presence of selected molecular alterations on primary tumour tissues and organoids | up to 5 years
  Concordance between the presence of selected molecular alterations on primary tumour tissues and organoids, frequencies will be reported and Cohen's Kappa will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Canzonieri, MD,PhD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS
Locations (1):
- Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS, Aviano, Pordenone, Italy